CLINICAL TRIAL: NCT03564197
Title: 18F-PD-L1 PET/CT to Predict Response to Nivolumab in Patients With NSCLC
Brief Title: 18F-PD-L1 PET/CT in Nivolumab Treated Patients With NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M17FNN; CA209-9XC (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-04-11; First posted 2018-06-20 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: NSCLC Stage IV
Keywords: EGFR WT; negative EML4-ALK fusion; eligible for first line chemo-immunotherapy, first line nivolumab/ipilimumab or 2nd line and beyond PD-(L)1 immunotherapy monotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Other): nivolumab containing treatment according to label
  Interventions: Other: 18F-PD-L1

INTERVENTIONS:
Other: 18F-PD-L1 — 18F-PD-L1 PET/CT scan
  Other Names: tracer

SUMMARY:
A multicenter single arm biomarker exploration and validation study. Eighty patients with NSCLC that are eligible for first line chemo-immunotherapy, first line nivolumab/ipilimumab or 2nd line and beyond PD-(L)1 immunotherapy monotherapy according to EMA label and national guidelines will be enrolled in this trial. All subjects will undergo a whole body 18F-PD-L1 PET/CT scan before start of nivolumab containing treatment. Patients will continue treatment until disease progression, withdrawal of patient consent or unacceptable toxicity.

DETAILED DESCRIPTION:
18F-PD-L1 PET/CT scan to predict durable reponse to nivolumab containing treatment in patients with NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of stage IV, EGFR WT and EML4-ALK fusion negative NSCLC. Mutational testing is not necessary in patients with squamous NSCLC.
2. Eligible for first line chemo-immunotherapy, first line nivolumab + ipilimumab or 2nd line and beyond PD-(L)1 immunotherapy monotherapy.
3. Be willing and able to provide written informed consent for the trial.
4. Be >= 18 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1.
6. Must provide tissue from a histological biopsy of a tumor lesion that is not radiated prior to biopsy and obtained after the last line of systemic therapy, to determine the actual PD-L1 status.
7. Have a performance status of 0-1 on the ECOG Performance Scale.
8. Demonstrate adequate hematologic and organ function, defined by the following laboratory results. All screening laboratory tests should be performed within 30 days prior to day 1 (PET imaging):

   * Absolute neutrophil count (ANC) ≥ 1500 cells/µL
   * WBC count ≥ 2000 cells/µL
   * Platelet count ≥ 100.000/µL
   * Hemoglobin ≥ 5.6 mmol/L
   * AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases are present)
   * Serum bilirubin ≤ 1.5 x ULN (except subjects with known Gilbert disease, who can have total bilirubin < 3.0 mg/dL)
   * Serum Creatinine ≤ 1.5 x ULN OR measured of calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 40 mL/min for subject with creatinine levels > 1.5 x ULN.

Exclusion Criteria:

1. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to day 1 (PET imaging). Inhaled or topical steroids, and adrenal replacement steroid >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
2. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
3. Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.

   * Note: Subjects with asymptomatic CNS metastases are allowed to enter the study.
   * Note: Subjects with previously treated brain metastases may participate provided they are clinically stable and not using steroids with > 10 mg daily prednisone equivalent for at least 7 days prior to trial treatment.
4. Has an active autoimmune disease requiring systemic steroid treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids.
5. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
6. Has an active infection requiring systemic therapy.
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
8. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks after the last dose of trial treatment.
10. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
11. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
12. Has known active Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival of >= 9 months | From date of registration until the date of progression-free survival >= 9 months (according to RECIST1.1)
  The outcome measures of 18F-PD-L1 PET/CT related to the progression-free survival at 9 months according to RECIST 1.1

SECONDARY OUTCOMES:
Progression Free Survival | From date of registration until the date of first documented progression assessed up to 5 months
  The outcome measures of 18F-PD-L1 PET/CT related to the date of the first documented tumor progression as determined by modified RECIST, or death due to any cause
Overall Survival | From date of registration until the date of death assessed up to 12 months
  The outcome measures of 18F-PD-L1 PET/CT related to the date of death due to any cause
Tumor and stromal PD-L1 IHC. | Through study completion, an average of 2 years
  Correlation between PD-L1 expression measured by 18F-PD-L1 PET/CT and PD-L1 expression measured by IHC

CONTACTS AND LOCATIONS:
Overall Officials: Joop de Langen, MD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek; Egbert Smit, MD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek
Locations (8):
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - MeanderMC, Amersfoort
  - VUmc, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - LUMC, Leiden
  - Medisch Centrum Haaglanden, The Hague
  - Antonius Ziekenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
to be decided